CLINICAL TRIAL: NCT01010022
Title: Examination of Safety and Efficacy of 6% Hydroxyethyl Starch 130/0.4 vs. 6% Hydroxyethyl Starch 70/0.5 in Patients Undergoing Orthopedic Surgery - a Double-blind, Parallel Group, Comparative, Multi-centre Phase III Study
Brief Title: Trial of 6% HES130/0.4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi Japan (Industry)
Responsible Party: Tsuneo Tsubaki, PhD, Pharm.D., Fresenius Kabi Japan K.K.
Organization: Fresenius Kabi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-13-02-JP
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Hypovolemia; Hemorrhage
Keywords: hypovolemia; surgical blood loss; orthopedic procedures; Treatment of reduced circulating blood volume (hypovolemia) including massive hemorrhage
MeSH Terms: conditions — Hypovolemia; Hemorrhage; Blood Loss, Surgical | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Up to 1000mL 6% hydroxyethyl starch 130/0.4 solution i.v., intra-operatively (from start of surgery until end of surgery)
  Interventions: Drug: 6% hydroxyethyl starch 130/0.4
- 2 (Active Comparator): Up to 1000mL 6% hydroxyethyl starch 70/0.5 (Salinhes®) solution i.v., intra-operatively (from start of surgery until end of surgery)
  Interventions: Drug: 6% hydroxyethyl starch 70/0.5 (Salinhes®)

INTERVENTIONS:
Drug: 6% hydroxyethyl starch 130/0.4 — Up to 1000mL 6% hydroxyethyl starch 130/0.4 solution i.v., intra-operatively (from start of surgery until end of surgery)
  Arms: 1
Drug: 6% hydroxyethyl starch 70/0.5 (Salinhes®) — Up to 1000mL 6% hydroxyethyl starch 70/0.5 (Salinhes®) solution i.v., intra-operatively (from start of surgery until end of surgery)
  Arms: 2

SUMMARY:
The study shall evaluate the efficacy and safety of two different hydroxyethyl starch solutions (artificial colloids 6% HES130/0.4 and 6% HES70/0.5, Salinhes®) for intra-operative therapy of hypovolemia and maintenance of circulating blood volume in patients undergoing orthopedic surgery. The primary efficacy endpoint will be the required volume of colloid solution infused from start until end of surgery. It is the aim of the clinical trial to demonstrate that comparable volumes of colloid solution are used between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an expected blood loss of ≥ 300 mL undergoing elective orthopedic surgery
* Patients with a body weight (BW) ≥ 50 kg

Exclusion Criteria:

* Known or suspected allergy to hydroxyethyl starch, including its ingredients (inclusive corn) and related drugs
* ASA classification ≥ IV
* Renal disease (serum creatinine ≥ 2mg/dL)
* Known bleeding disorders
* Congestive heart failure
* Fluid overload
* Intracranial bleeding
* Severe hypernatremia
* Severe hyperchloremia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Volume of colloid solution infused during investigational period (= intra-operatively) | Intra-operatively

SECONDARY OUTCOMES:
Fluid input | From immediately before induction of anesthesia until 48 hours after end of surgery
Fluid output | From immediately before induction of anesthesia until 48 hours after end of surgery
Fluid balance | From immediately before induction of anesthesia until 48 hours after end of surgery
Hemodynamics | From immediately before induction of anesthesia until 48 hours after end of surgery
Co-administration of vasoactive drugs | From enrolment until 48 hours after end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Akiyoshi Namiki, MD, PhD, Study Chair — Emeritus Professor, Sapporo Medical University
Locations (7):
- Japan (7):
  - Sapporo Medical University, School of Medicine, Sapporo, Hokkaido
  - Kyushu University, Graduate School of Medical Sciences, Fukuoka
  - Kobe University Graduate School of Medicine, Kobe
  - Okayama University, Okayama
  - Osaka University Graduate School of Medicine, Osaka
  - Keio University School of Medicine, Tokyo
  - Tokyo Women's Medical University, Tokyo